CLINICAL TRIAL: NCT00501410
Title: Dual Inhibition of EGFR and c-Src by Cetuximab and Dasatinib Combined With FOLFOX Chemotherapy in Metastatic Colorectal Cancer (CA180048)
Brief Title: FOLFOX Chemotherapy Regimen (5-FU, Leucovorin, Oxaliplatin) in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0842; NCI-2015-01568 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Dual Inhibition of EGFR; FOLFOX Chemotherapy; 5-FU; Cetuximab; Dasatinib; Leucovorin; Oxaliplatin; 5-Fluorouracil; BMS-354825; Eloxatin; Sprycel; C225; Erbitux; IMC-C225; Adrucil; Efudex; Folinic Acid
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Cetuximab; Dasatinib; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FOLFOX + Dasatinib + Cetuximab (Experimental): 5-FU 2400 mg/m^2 by vein over 46 Hours On Days 1 & 2. Cetuximab initial dose = 400 mg/m^2 by vein, then 250 mg/m^2 Weekly On Days 1 & 8. Dasatinib 100 mg by mouth daily on days 1-14. Leucovorin 400 mg/m^2 by vein on day 1. Oxaliplatin 85 mg/m^2 by vein on day 1.
  Interventions: Drug: 5-FU; Drug: Cetuximab; Drug: Dasatinib; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5-FU — 2400 mg/m^2 by vein over 46 Hours On Days 1 & 2.
  Other Names: 5-Fluorouracil
Drug: Cetuximab — Initial Dose = 400 mg/m^2 by vein, then 250 mg/m^2 Weekly On Days 1 & 8
Drug: Dasatinib — Starting dose level: 100 mg by mouth daily on days 1-14.
  Other Names: BMS-354825
Drug: Leucovorin — 400 mg/m^2 by vein on day 1.
  Other Names: Folinic Acid
Drug: Oxaliplatin — 85 mg/m^2 by vein on day 1.
  Other Names: Eloxatin

SUMMARY:
The goal of the Phase I part of this clinical research study is to find the highest tolerable dose of a combination of dasatinib, cetuximab, and FOLFOX (5-fluorouracil [5-FU], leucovorin [LV], and Eloxatin [oxaliplatin]) that can be given to patients with metastatic colorectal cancer. The safety of these drugs in combination will also be studied.

The goal of the Phase II part of this clinical research study is to learn if dasatinib given in combination with FOLFOX with or without cetuximab can help to control metastatic colorectal cancer.

DETAILED DESCRIPTION:
Cetuximab is a drug designed to block the activity of EGFR, a protein on the surface of some tumor cells that may cause the cells to grow. Blocking EGFR may stop or slow the growth of tumor cells. Dasatinib is a drug that inhibits a protein called c-Src. High levels of c-Src may make it harder for chemotherapy to work against the cancer. If dasatinib can inhibit c-Src, the chemotherapy may be more effective against the cancer. FOLFOX is a drug combination frequently used to treat colon or rectal cancer that has spread to other parts of the body. FOLFOX is designed to kill rapidly dividing cells by preventing DNA (the genetic material of cells) from duplicating.

Kirsten Rat Sarcoma (KRAS) Testing:

Recent studies have found that cetuximab, when given alone or in combination with other chemotherapy drugs, was not effective when given to patients with colorectal cancer that had a KRAS gene mutation.

If you take part in the Phase I part of this study, your tumor tissue from a previous biopsy or surgery will be used to test for KRAS mutation. If you have the KRAS gene mutation, you will not take part in this study.

If you take part in the Phase II part of this study, your tumor tissue from a previous biopsy or surgery will be used to test for KRAS mutation. If you have the KRAS gene mutation, you may take part in the study but you will not receive cetuximab.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group (Phase I or Phase II) based on when you join this study.

If you are enrolled in the Phase I portion, the dose of dasatinib you will receive will depend on when you joined the study. Three (3) to 6 participants will be entered at each dose level. Each new group of participants will receive a higher dose, until the highest tolerable dose is found. Once the highest tolerable dose is found, 12 participants will be enrolled at that dose level. Your doctor will tell you what dose level you will be receiving and how this dose compares to the doses other participants have received. The starting dose of cetuximab and FOLFOX will be the same for all participants. The dose of dasatinib will be increased with the next group of 3-6 participants. Every 14 days is considered 1 study "cycle".

If you are enrolled in the Phase II portion, you will receive the dose of dasatinib found to be best tolerated in the Phase I portion. You will also receive FOLFOX. If you do not have the KRAS gene mutation, you will also receive cetuximab. Every 14 days is considered 1 study "cycle".

Central Venous Catheter (CVC) Placement:

Before receiving the study drugs, you will have a CVC placed. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

Study Drug Administration:

You will take dasatinib by mouth once a day, every day during this study. Your study doctor and research nurse will tell you how many pills you will take. Dasatinib should be taken at the same time each day, with or without meals. If you miss a dose of dasatinib, you should not double the next dose. It is important to take dasatinib with water, and not fruit juices. You should not drink grapefruit juice or eat grapefruit while you are on this study. Dasatinib should not be touched by children, pregnant women, or women who are breastfeeding. If a caregiver must handle the drug, a protective glove should be worn.

While you are taking dasatinib, you will be given a drug diary. In this diary, you will write down the date, the time, and the number of dasatinib tablets taken. Certain drugs and herbal supplements may not be taken while you are receiving dasatinib. These drugs could affect how your body breaks down dasatinib, which could have a bad effect on you. Your doctor will give you a list of drugs and herbal supplements that you must not take while on this study. You must tell your doctor before taking any new drugs while on this study.

On Day 1 of every cycle, you will receive oxaliplatin and LV through the CVC over about 2 hours. On Day 1, you will receive 5-FU through a portable pump for the next 46 hours. If you are receiving cetuximab in the Phase I portion of the study, you will receive it on Days 1 and 8 through the CVC over about 2 hours. If you are receiving cetuximab in the Phase II portion of the study, you will receive it on Day 1 through the CVC over about 2 hours.

Study Visits for Phase I:

If you are enrolled at the highest tolerable dose level, you will have 2 core liver biopsies. The liver tissue will be studied to learn the effect of the study drugs on stopping the protein c-Src. You will have 2 liver biopsies collected. The first liver biopsy will be collected before you start the study drugs, and the second will be performed in either Cycle 2 or 3. Before the liver biopsy, you will receive fluids and drugs for relaxation and/or pain through an needle in your arm or hand. You will be awake during the biopsy. A radiologist will find the tumor in the liver with the help of radiographic imaging procedures such as an ultrasound or CT scan. Your skin around this area will be cleansed, and a local anesthetic will be given. A long, hollow needle will be inserted through the skin into the liver tumor, and a tissue sample(s) will be taken.

On Day 8, blood (about 1-2 tablespoons) will be drawn for routine tests.

You will have extra blood samples drawn (1 tablespoon each time) before receiving the study drugs and on Day 8 of Cycles 2 and 4. This blood will be drawn at the same time as your routine blood tests are drawn. These blood samples will be used to develop tests that may help doctors be able to predict who will best benefit from dasatinib.

If you are enrolled in the group that receives the highest tolerable dose level, the Day 8 blood draw during cycle 2 will not be performed. Instead, blood will be collected at the time of the liver biopsy that is to be performed between Days 8-14 of cycle 2 or 3 about 2 to 6 hours after taking the daily dose of dasatinib.

Study Visits for Phase II:

You will have extra blood samples drawn (1 tablespoon each time) before receiving the study drugs and at the end of every 4 cycles. This blood will be drawn at the same time as your routine blood tests are drawn. These blood samples will be used to develop tests that may help doctors be able to predict who will best benefit from dasatinib.

Before the start of each new cycle and when you stop study treatment, you will be asked to complete a questionnaire about any symptoms you may be experiencing. The questionnaire will take up to 5 minutes to complete.

Once you stop receiving study drugs, the study team will contact you by telephone every 3 months to check how you are doing. Each phone call will take about 5 minutes.

Phase I and Phase II:

Before each new cycle, you will be asked questions about any side effects you may have had. At each visit, it is important to tell the study staff about any drugs you are currently taking. You will have a physical exam, including measurement of your vital signs and weight. You will have a performance status evaluation. Blood (about 1-2 tablespoons) will be drawn for routine tests.

Women who are able to become pregnant will have a blood or urine pregnancy test every month.

If you experience severe side effects, the study drugs may be delayed, stopped, or you may receive smaller doses of the drugs.

You may remain on this study for as long as you are benefiting. You will be taken off this study if the disease gets worse or intolerable side effects occur.

Once you are off-study, you will have an end-of-study visit. At this visit, blood (about 3 tablespoons) will be collected for routine tests. You will be asked questions about any side effects you may have had and about any drugs you are currently taking. You will have a physical exam, including measurement of your vital signs and weight. You will have a performance status evaluation. If not performed recently, you will have a CT scan or MRI scan of your chest, abdomen and pelvis to check the status of the disease. If you are having side effects after you stop receiving the study drugs, you will be contacted by phone to check how you are feeling, or you will have follow-up visits until the side effects have gone away.

This is an investigational study. Dasatinib is FDA approved for the treatment of leukemia. Its use in this study, for this disease, is considered to be investigational. Cetuximab, 5-FU, LV, and oxaliplatin are all FDA approved and commercially available for the treatment of colorectal cancer. Up to 83 patients will take part in this study. All patients will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically or cytologically confirmed colorectal adenocarcinoma with metastatic disease documented on diagnostic imaging studies
2. Phase IB: Patient must have wild type KRAS.
3. Phase IB: For the expansion cohort, only patients with liver metastases >/= 2.0 cm amenable to percutaneous CT or U/S guided biopsy and who agree to having 2 liver biopsies done are eligible.
4. Phase II: Patient must have known KRAS (exon 1, codon 12, 13) or sufficient available tumor tissue from the primary tumor or metastatic site for KRAS mutation analysis [Phase II only].
5. Patient must have previously progressed on systemic therapy for metastatic colorectal cancer, with no limit on the number of prior regimens. For patients in the Phase II cohort, they must have progressed on 5-FU or capecitabine and oxaliplatin [patients with KRAS mutated tumors], and either cetuximab or panitumumab [patients with KRAS wild type tumors].
6. (Continued from # 5) The following criteria must be met for progression. • Baseline imaging was performed 1 month or less prior to starting regimen. • Average treatment intensity (number of cycles received/number of cycles anticipated in absence of delays) of greater than 70%. • Restaging study demonstrating progression 6 weeks or less from last dose of oxaliplatin and EGFR inhibitor (if applicable). • Progression may be by RECIST criteria or, with PI approval, clinical progression.
7. Written informed consent obtained
8. Age >/= 18 years to provide a uniform oncologic phenotype of adult-onset colorectal cancer.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Appendix E)
10. Patients must have adequate organ and marrow function defined as: absolute neutrophil count (ANC) >/= 1,500/mm^3; platelets >/= 100,000/ mm^3; hemoglobin >/= 9 gm/dL (may be transfused to maintain or exceed this level); total bilirubin </= 1.5 mg/dL; AST (SGOT)/ALT(SGPT) </= 2.5 times institution's upper limit of normal (IULN), or </= 5 times IULN if known liver metastases; · Creatinine clearance > 60mL/min using Cockcroft-Gault formula.
11. Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the start of study medications. Childbearing potential is defined as a woman who is not post-menopausal for 12 months or longer or is not surgically sterile. Patients must agree to practice acceptable contraceptive methods as outlined in the protocol.

Exclusion Criteria:

1. Recent (within 4 weeks of the first infusion of study drugs on this study), or planned participation in another experimental therapeutic drug study. Patients who have had any systemic chemotherapy, radiotherapy, or major surgery within 21 days prior to the first infusion of study drugs.
2. Patients who have not recovered to </= grade 2 for neuropathy or </= grade 1 for other side effects due to prior treatment.
3. Patients with radiographic evidence of pleural effusions in the last 30 days prior to enrollment.
4. Patients with known brain metastases because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
5. Female patients who are pregnant or lactating or men and women of reproductive potential not willing to employ an effective method of birth control during treatment and for 3 weeks after discontinuing study treatment
6. Patients with known dihydropyrimidine dehydrogenase deficiency.
7. Patients with a history of significant bleeding disorder unrelated to cancer, including: Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease); Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
8. Patients currently taking the following drugs that are generally accepted to have a risk of causing Torsades de Pointes:haloperidol, methadone, amiodarone, sotalol, erythromycins, clarithromycin cisapride, chlorpromazine, bepridil, droperidol, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine, quinidine, procainamide, disopyramide, ibutilide, dofetilide. Subjects who have discontinued any of these medications must have a wash-out of at least 5 days (or 14 days for amiodarone) prior to the first dose of dasatinib.
9. Patients with wild type KRAS tumors with a history of allergic reactions attributed to cetuximab, oxaliplatin, 5-FU, capecitabine, or leucovorin that, previously, have not been adequately prevented with premedications.
10. Current use of full-dose warfarin (except as required to maintain patency of preexisting, permanent indwelling IV catheters). For subjects receiving warfarin for catheter patency, international normalized ratio (INR) should be < 1.5.
11. Current or recent (<2 week) use of aspirin (at a dose greater than 81 mg/day) or clopidogrel.
12. Diagnosed or suspected congenital long QT syndrome
13. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes).
14. Previous allergic reaction to a human monoclonal antibody.
15. Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec) on both the Fridericia [QTc = QT/RR^1/3] and Bazett's [QTc = QT/sqrtRR] correction. Bazett's correction is calculated automatically by institutional EKG machines
16. Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study: Uncontrolled high blood pressure (systolic blood pressure >/= 140 and diastolic blood pressure >/= 90), history of labile hypertension, or history of poor compliance with an antihypertensive regimen. Unstable angina or stable angina markedly limiting ordinary physical activity. (Angina occurs on walking one to two blocks on the level and climbing one flight of stairs in normal conditions and at a normal pace) .
17. Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study: New York Heart Association (NYHA) >/= grade 2 congestive heart failure; Myocardial infarction within 6 months of study enrollment; History of stroke within 6 months of study enrollment; Unstable symptomatic arrhythmia requiring medication (Patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal SVT are eligible); Clinically significant peripheral vascular disease; Uncontrolled diabetes; Serious active or uncontrolled infection
18. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of a study drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
19. Inability to take oral medications.
20. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-04-23 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Dasatinib, Cetuximab and FOLFOX | 2 Week Cycles
  If 2 or more out of the 6 patients in the cohort have dose limiting toxicity (DLT) then the prior dose level is the MTD.

SECONDARY OUTCOMES:
Response-Rate of Dasatinib and Modified FOLFOX6 With or Without Cetuximab | After 4, 14 day cycles
  Response and progression evaluated using a modification of the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000]. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria. Duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org